CLINICAL TRIAL: NCT01176682
Title: European Real Life Study on NSAIDs Treated Patients With Osteoarthritis (OA), Rheumatoid Arthritis (RA) and Ankylosing Spondylitis (AS): Assessment of Pain Relieve, Gastrointestinal (GI) Symptoms, Adherence and Health Resource Consumption
Brief Title: Observational Study on Non-steroid Anti-inflammatory Drugs (NSAIDs) Treated Patients With Arthritic Disorder
Acronym: EVIDENCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GEU-DUM-2010/1
Record Dates: First submitted 2010-07-30; First posted 2010-08-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: NSAID-treated patients; gastrointestinal events; Non-steroid anti-inflammatory drug (NSAID); Gastrointestinal events (GI events); Proton Pump Inhibitors (PPI)
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult patients treated with NSAID therapy for diagnosed OA, RA or AS, and with GI risk factors

SUMMARY:
The aim of this study is to find out how patients with osteoarthritis, rheumatoid arthritis and ankylosing spondylitis receiving NSAID-therapy are treated and managed by their doctor in usual clinical practice, how patients comply with their treatment and how satisfied they are with their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of arthritic disorder (osteoarthritis, rheumatoid arthritis or ankylosing spondylitis)
* Already receiving NSAID treatment at enrolment visit

Exclusion Criteria:

* Inability to complete the study related questionnaires
* Current participation in any interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with NSAID therapy for diagnosed OA, RA or AS, and with GI risk factors. The patients will be asked to participate by their treating doctors at GP centres, specialist centres or hospitals.
  Participating investigators will belong to a variety of centres representing the reality of how and where these patients are managed in each country.
Sampling Method: Non-Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The incidence of selected GI events, classified as "symptomatic" or "complicated" GI events. Reported by the patients at the follow-up visits. | Time from NSAID treatment prescription to first diagnosis of the GI event for each patient will be registered. Each patient will be followed up for 6 months.

SECONDARY OUTCOMES:
Number of health care visits and days of hospitalisation (health care consumption) related to arthritic disorder and/or GI events as reported by the patients at the follow-up visits. | Health care consumption accumulated over the 6 months study period will be registered.
Quality of life assessed by EuroQol-5 Dimension (EQ-5D) at baseline and the follow-up visits. Measure how selected GI events impact the EQ-5D score. | Measurements at baseline, 3 months and 6 months
Adherence with NSAIDs and proton pump inhibitors (PPI) measured by Morisky-Green-Levine Medication Assessment Scale (MMAS) at baseline and follow-up visits. | Measurements at baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Nuevo, MSc, Study Director — Medical Department.AstraZeneca Spain
Locations (244):
- Belgium (43):
  - Research Site, Alsemberg
  - Research Site, Anthée
  - Research Site, Baisy-Thy
  - Research Site, Blankenberge
  - Research Site, Bois-de-Villers
  - Research Site, Brussels
  - Research Site, Champion
  - Research Site, Chênée
  - Research Site, Dour
  - Research Site, Ecaussinnes
  - Research Site, Fosses-la-Ville
  - Research Site, Geel
  - Research Site, Genly
  - Research Site, Godinne
  - Research Site, Gozée
  - Research Site, Gribomont
  - Research Site, Halen
  - Research Site, Ham-sur-Heure-Nalinnes
  - Research Site, Hasselt
  - Research Site, Hove
  - Research Site, Kraainem
  - Research Site, Libramont-Chevigny
  - Research Site, Linkebeek
  - Research Site, Lommel
  - Research Site, Marchovelette
  - Research Site, Melsbroek
  - Research Site, Moerkerke-Damme
  - Research Site, Mont-sur-Marchienne
  - Research Site, Mouscron
  - Research Site, Natoye
  - Research Site, Oostham
  - Research Site, Retie
  - Research Site, Ronquières
  - Research Site, Rumst
  - Research Site, Saint-Ghislain
  - Research Site, Seraing
  - Research Site, Sint-Amands
  - Research Site, Thuillies
  - Research Site, Tremelo
  - Research Site, Turnhout
  - Research Site, Veurne
  - Research Site, Vilvoorde
  - Research Site, Zoersel
- France (46):
  - Research Site, Arches
  - Research Site, Art-sur-Meurthe
  - Research Site, Aubagne
  - Research Site, Banyuls de la Marenda
  - Research Site, Bassussarry
  - Research Site, Cappelle-en-Pévèle
  - Research Site, Castets
  - Research Site, Champagnole
  - Research Site, Charvieu-Chavagneux
  - Research Site, Colmar
  - Research Site, Couzeix
  - Research Site, Firminy
  - Research Site, Fleury-sur-Orne
  - Research Site, Gallardon
  - Research Site, Gelles
  - Research Site, La Motte-Servolex
  - Research Site, Lambersart
  - Research Site, Le Bois-dOingt
  - Research Site, Le Bouscat
  - Research Site, Le Cannet
  - Research Site, Le Pontet
  - Research Site, Le Russey
  - Research Site, Lembach
  - Research Site, Marles-les-Mines
  - Research Site, Marseille
  - Research Site, Mensignac
  - Research Site, Moreuil
  - Research Site, Mourmelon-le-Petit
  - Research Site, Narbonne
  - Research Site, Neuilly-lès-Dijon
  - Research Site, Noyon
  - Research Site, Paris
  - Research Site, Pisany
  - Research Site, Puyricard
  - Research Site, Roissy-en-France
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Estève
  - Research Site, Saint-Martin-de-Crau
  - Research Site, Salles
  - Research Site, Sonchamp
  - Research Site, Ste Fortunade
  - Research Site, Ste Severe Sur Indre
  - Research Site, Toulon
  - Research Site, Villejuif
  - Research Site, Voisins-le-Bretonneux
  - Research Site, Waziers
- Germany (23):
  - Research Site, Aiterhofen
  - Research Site, Bad Salzuflen
  - Research Site, Bergkamen
  - Research Site, Blankenhain
  - Research Site, Bockenem
  - Research Site, Cologne
  - Research Site, Deggingen
  - Research Site, Essen
  - Research Site, Gortringen
  - Research Site, Hamburg
  - Research Site, Lengerich
  - Research Site, Lenne
  - Research Site, Ludwigshafen
  - Research Site, Offenbach
  - Research Site, Potsdam
  - Research Site, Reinfeld
  - Research Site, Remscheid
  - Research Site, Rodgau
  - Research Site, Spaichingen
  - Research Site, Stockach
  - Research Site, Wangen
  - Research Site, Wardenburg
  - Research Site, Weinheim
- Greece (12):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Drama
  - Research Site, Florina
  - Research Site, Heraklion
  - Research Site, Karditsa
  - Research Site, Kastoria
  - Research Site, Kozani
  - Research Site, Serres
  - Research Site, Thessaloniki
  - Research Site, Trikala
  - Research Site, Xánthi
- Italy (3):
  - Research Site, Salerno
  - Research Site, Varese
  - Research Site, Viareggio
- Netherlands (19):
  - Research Site, Amsterdam
  - Research Site, Andijk
  - Research Site, Bennebroek
  - Research Site, Dordrecht
  - Research Site, Ermelo
  - Research Site, Lichtenvoorde
  - Research Site, Lieshout
  - Research Site, Losser
  - Research Site, Nijmegen
  - Research Site, Nijverdal
  - Research Site, Rijswijk
  - Research Site, Rilland
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, Soerendonk
  - Research Site, Spijkenisse
  - Research Site, The Hague
  - Research Site, Volendam
  - Research Site, Woerden
- Norway (17):
  - Research Site, Årnes
  - Research Site, Baverbru
  - Research Site, Eydehavn
  - Research Site, Fornebu
  - Research Site, Frogner
  - Research Site, Hurdal
  - Research Site, Kirkenær
  - Research Site, Lierskogen
  - Research Site, Lillestrøm
  - Research Site, Mosterhamn
  - Research Site, Nordlenangen
  - Research Site, Oslo
  - Research Site, Rodal
  - Research Site, Skien
  - Research Site, Strømmen
  - Research Site, Svelvik
  - Research Site, Tanager
- Spain (7):
  - Research Site, Campotéjar
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Málaga
  - Research Site, Nigrán
  - Research Site, Tomiño
  - Research Site, Vigo
- Sweden (10):
  - Research Site, Dalby
  - Research Site, Gothenburg
  - Research Site, Kristianstad
  - Research Site, Lidingö
  - Research Site, Limhamn
  - Research Site, Pitee
  - Research Site, Skanör
  - Research Site, Stockholm
  - Research Site, Vonnes
  - Research Site, Ystad
- Switzerland (14):
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Brittnau
  - Research Site, Buchs
  - Research Site, Chiasso
  - Research Site, Chur
  - Research Site, Egg Bei Zurich
  - Research Site, Ilanz
  - Research Site, Oberwil
  - Research Site, Sankt Gallen
  - Research Site, Sarmenstorf
  - Research Site, Schiers
  - Research Site, Wallisellen
  - Research Site, Zurich
- Turkey (Türkiye) (17):
  - Research Site, ?stanbul
  - Research Site, ?zmir
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Ayd?n
  - Research Site, Bursa
  - Research Site, Diyarbak?r
  - Research Site, Elaz??
  - Research Site, Erzurum
  - Research Site, Eski?ehir
  - Research Site, Isparta
  - Research Site, Kastamonu
  - Research Site, Kayseri
  - Research Site, Konya
  - Research Site, Manisa
  - Research Site, Trabzon
  - Research Site, Van
- United Kingdom (33):
  - Research Site, Addlestone, Surrey
  - Research Site, Ashford, Middlesex
  - Research Site, Aston Clinton, Bucks
  - Research Site, Atherstone, Warwickshire
  - Research Site, Bangor, Northern Ireland
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bradford-On-Avon, Wiltshire
  - Research Site, Cookstown, Northern Ireland
  - Research Site, Coventry
  - Research Site, Crawley, West Sussex
  - Research Site, Cumbernauld
  - Research Site, Frome, Wiltshire
  - Research Site, Glasgow
  - Research Site, Harrow, Middlesex
  - Research Site, High Valleyfield, Fife
  - Research Site, Irvine
  - Research Site, Maidenhead
  - Research Site, Motherwell
  - Research Site, New Stevenson
  - Research Site, Newcastle upon Tyne
  - Research Site, Pound Hill, Crawley
  - Research Site, Randalstown
  - Research Site, Royal Leamington Spa
  - Research Site, Sneinton, Nottingham
  - Research Site, Stevenage
  - Research Site, Titchfield
  - Research Site, Trowbridge
  - Research Site, Warminster
  - Research Site, Watford
  - Research Site, Wellingborough
  - Research Site, Woolpit, Bury Saint Edmonds

REFERENCES:
- [Derived] Lanas A, Boers M, Nuevo J. Gastrointestinal events in at-risk patients starting non-steroidal anti-inflammatory drugs (NSAIDs) for rheumatic diseases: the EVIDENCE study of European routine practice. Ann Rheum Dis. 2015 Apr;74(4):675-81. doi: 10.1136/annrheumdis-2013-204155. Epub 2013 Dec 18. PMID 24351518